CLINICAL TRIAL: NCT06826417
Title: Pain, Anxiety and Anesthetic Satisfaction for Patient With Different State Anxiety Underwent Cataract Surgery With Topical Anesthesia
Brief Title: Anxiety and Surgery Satisfaction for Cataract Patient With Different State Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 202302067MINB
Record Dates: First submitted 2024-12-12; First posted 2025-02-14 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Oral Anxiolytic; Phacoemulsification; Cataract Surgery; Satisfaction Survey; State Anxiety
Keywords: Oral anxiolytic; Phacoemulsification; Cataract surgery; Satisfaction survey; State Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Alprazolam

STUDY DESIGN:
Intervention Model Description: Double-blind randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xanax (Experimental)
  Interventions: Drug: Xanax
- Placebo (Placebo Comparator)
  Interventions: Other: placebo tablets

INTERVENTIONS:
Drug: Xanax — double-blind randomized controlled clinical trial: in a double-blind manner, to receive Xanax
  Arms: Xanax
Other: placebo tablets — double-blind randomized controlled clinical trial: in a double-blind manner, to receive a placebo (identical in appearance to Xanax but without any active effects)
  Other Names: placebo
  Arms: Placebo

SUMMARY:
This study aims to explore the effects of anxiety traits on pain, anxiety, and anesthesia satisfaction in patients undergoing cataract surgery under topical anesthesia. On the day of recruitment, patients will complete the BAI, STAI-S, and STAI-T anxiety questionnaires to assess baseline anxiety levels. Thirty minutes before the surgery, patients will be randomly assigned, in a double-blind manner, to receive either Xanax or a placebo and will retake the BAI, STAI-S, and STAI-T questionnaires. After the surgery, patients' pain levels and anesthesia satisfaction will be evaluated, with the pain scale and satisfaction survey repeated the following day. The results will analyze the relationship between anxiety traits and pharmacological interventions on the surgical experience, aiming to optimize surgical procedures and improve overall patient comfort.

DETAILED DESCRIPTION:
BACKGROUNDS Nowadays, phacoemulsification for cataract treatment is the most common surgical procedure performed and anesthetics procedure has been shifted from retrobulbar or peribulbar anesthesia to topical anesthesia (TA). Phacoemulsification under TA is proved to be a safe and low risk procedure with the incidence of adverse events requiring medical emergency team interventions to be 0.04%. However, it is not uncommon that patients can suffer from pain, anxiety and unpleasant visual sensation during this procedure. Complementary sedation has long been thought to alleviate the anxiety and pain of the patient during surgery with local anesthesia. Studies revealed that approximate one fourth of the patients underwent phacoemulsification under TA or retrobulbar anesthesia requested additional intravenous sedation of midazolam. However, the intravenous sedation, such as midazolam, propofol, or etomidate, increase the risk of additional anesthetic complications of heart rate, blood pressure, body temperature, and nausea, and therefore, anesthesia monitoring was mandatory during the surgery.

Compared with intravenous sedation, oral sedation is less costly and less invasive. Studies with different oral sedation agents revealed different effect. In the study of 41 patients serving themselves as control, patients reported more pain and photophobia in the surgery with TA alone than the other with midazolam syrup and oral transmucosal fentanyl citrate. However, two studies comparing oral diazepam or triazolam with intravenous midazolam showed similar rate of anxiety and pain or noninferior satisfaction. Moreover, the randomized control trial containing 50 procedures in each groups revealed that patients received TA alone during phacoemulsification reported similar pain or anxiety level to those received complementary intravenous midazolam.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years old.
2. Patients diagnosed with cataracts.
3. Scheduled for cataract surgery with phacoemulsification and intraocular lens implantation under surface anesthesia at National Taiwan University Hospital.
4. No adverse reactions to oral anti-anxiety medication (XANAX).

Exclusion Criteria:

1. Presence of any contraindications for surgery before the procedure.
2. Presence of any contraindications for medication before the procedure.
3. Inability to provide clear and complete answers to relevant questionnaires, or expression of no preoperative anxiety during the outpatient visit, or scores below 21 on the STAI-S or STAI-T assessment.
4. Regular use of anti-anxiety medications, sleeping pills, or analgesics before the procedure.
5. Pregnancy or breastfeeding during the preoperative period.
6. Severe corneal diseases, overripe cataracts, small pupils, or lens dislocation leading to difficulties in conventional surgery.
7. Patients under surface anesthesia who cannot fully cooperate with the surgical procedure.
8. Pregnant or uncertain pregnancy status (women under 55 years old to be verbally asked by research team members).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2026-09-11 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Beck Anxiety Inventory (BAI) | 1-3 months
  The Beck Anxiety Inventory (BAI) is a psychological scale specifically designed to assess symptoms of anxiety. The Chinese version has been translated and adapted for Chinese-speaking users. The inventory consists of 21 items covering physiological and cognitive anxiety symptoms, such as palpitations, breathlessness, and tension. Each item is rated on a 4-point scale (0 to 3) based on the frequency or severity of symptoms, with a total score range of 0 to 63. Higher scores indicate more severe anxiety. The BAI demonstrates strong reliability and validity, making it suitable for clinical diagnosis, psychological assessment, and research purposes. It helps clinicians and researchers quickly understand an individual's anxiety levels and evaluate intervention effectiveness.
State-Trait Anxiety Inventory (STAI-S / STAI-T) | 1-3 months
  The State-Trait Anxiety Inventory (STAI) is a psychological assessment tool designed to measure anxiety levels, focusing on state anxiety (SA) and trait anxiety (TA). The Chinese version has been translated and culturally adapted for Chinese-speaking users. The inventory comprises 40 items, with 20 items assessing state anxiety and 20 items assessing trait anxiety. Each item is rated on a 4-point scale (1 to 4), resulting in a total score range of 20 to 80 for both SA and TA. Higher scores indicate more severe anxiety. The STAI is widely recognized for its strong reliability and validity, making it suitable for clinical diagnosis, psychological assessment, and research purposes. It is particularly valuable in evaluating the effectiveness of interventions and understanding anxiety characteristics and trends across different populations.
Cataract Surgery Records: Surgical Procedure | 1 days
  Anesthesia Type: Peribulbar, Topicalanesthesia Incision Area: Corneal, Limbal, Scleral. Incision Location: O'clock position. Cumulative Dissipated Energy (CDE): % / second. Total Surgical Time: Minutes. Phacoemulsifi cation Technique: Phaco-chop, Stop and chop, Divide and conquer. IOL Type:Toric, Non-toric. Capsular Tension Ring (CTR) Use: Yes, No. Suture Presence: Yes, No. Zonular Laxity: Yes, No. Degree of Fixation Loss: Perfect, Fair, Not cooperative, Severedeviation. Number of Abnormal Head or Body Movements. Surgical Complications:Capsular rupture, Vitreous loss, Hyphema, Iris prolapse, Others (specify).
Cataract Surgery Records: Surgical Procedure (Intraoperative Monitoring) | 1 days
  Oxygen saturation (%).
Cataract Surgery Records: Surgical Procedure (Intraoperative Monitoring) | 1 days
  Blood pressure (mmHg).
Cataract Surgery Records: Surgical Procedure (Intraoperative Monitoring) | 1 days
  Heart rate (bpm).
Cataract Surgery Records: Pain Scale | 1 days
  Surgical Outcome: Initial outcomes immediately after surgery, including corneal clarity, IOL positioning, and patient reaction. Complication Management: Actions taken to address any intraoperative complications, such as hemostatic measures or additional medication. Pain Assessment: Documentation of immediate postoperative pain levels and pain management interventions.
Cataract Surgery Records: Anesthesia Satisfaction Rating Scale | 1 days
  The anesthesia satisfaction rating scale evaluates patients' satisfaction with the anesthesia experience during surgical procedures, focusing on factors such as pain management, comfort, and communication with the anesthesia team. The scales typically use a numerical rating system, such as a 10-point scale, where higher scores indicate greater satisfaction. These tools are simple and effective for assessing patients' perspectives on specific aspects of their care. The results are valuable for optimizing clinical procedures, improving patient experiences, and enhancing the quality of medical services.
Postoperative Follow-Up | 1 days
  Bulbar Injection: 0, 1, 2, 3, 4. Anterior Chamber Reaction (AC Reaction): 0, 1, 2, 3,4. Corneal Edema: 0, 1, 2, 3, 4. Intraocular Pressure (mmHg) (IOP): ≤21, >21. bulbar injection(0 to 4 +) (0) no injection; (1) very slight; (2) slight; (3) moderate; (4) severe.
  Anterior chamberreaction (cell 0 to 4+) in a 1 x 1 mm slit-lamp beam (0) No cells; (1+) 5-10 cells ; (2+)11-20 cells ;(3+) 21-50 cells ; (4+) >50 cells.
Postoperative Follow-Up (Postoperative Symptoms) | 1 days
  None; Fatigue; Ataxia; Dizziness; Headache; Urinary retention; Amnesia; Muscle weakness; Nausea; Confusion; Disorientation; Restlessness; Others (specify).
Postoperative Satisfaction Pain Scale | 1 days
  The pain scale is a tool for assessing patients' subjective perceptions of pain, widely used in clinical and research settings. It typically employs numerical ratings (e.g., 0-10) or a Visual Analog Scale (VAS), where 0 represents no pain and 10 represents the most severe pain. Patients select a score based on their experience, quantifying their pain levels in a straightforward manner. This tool is commonly used in postoperative, chronic pain, or acute pain management, helping healthcare providers quickly understand patients' pain conditions and adjust treatment plans accordingly. With its simplicity and high reliability, the pain scale is an essential standardized evaluation tool in the medical field.
Postoperative Satisfaction Rating Scale | 1 days
  The postoperative satisfaction rating scale assesses overall satisfaction with the surgical experience, including pain relief, medical care, and service quality. The scales typically use a numerical rating system, such as a 10-point scale, where higher scores indicate greater satisfaction. These tools are simple and effective for assessing patients' perspectives on specific aspects of their care. The results are valuable for optimizing clinical procedures, improving patient experiences, and enhancing the quality of medical services.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided